CLINICAL TRIAL: NCT05642364
Title: Positive Psychological Intervention Delivered Using Virtual Reality in Hemodialysis Patients With Comorbid Depression: Randomized Controlled Trial Assessing Feasibility and Efficacy Testing
Brief Title: Virtual Reality in Hemodialysis to Improve Psychological Well-being
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northwestern University (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Rosalba Hernandez, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01DK129594 (NIH); 5R01DK129594 (NIH)
Record Dates: First submitted 2022-06-13; First posted 2022-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: End Stage Kidney Disease; Depressive Symptoms
Keywords: Positive psychological intervention; Positive emotion; Virtual reality; Psychotherapy; Technology; Head-mounted display
MeSH Terms: conditions — Kidney Failure, Chronic; Depression

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled trial, inclusive of treatment group and attention-control condition
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will both receive virtual reality exposure, specifically the treatment condition will receive a 5-week VR-based positive psychological intervention and the control arm will be exposed to 2-dimensional wildlife footage and nature-based settings with inert music. The outcome assessor will not be aware of trial arm assignment and will not have interaction with patient enrollees in any other capacity of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Treatment (Experimental): VR-delivered JovialityTM Sessions: Treatment Group. Participants will interact with a newly-developed VR environment over a 5-week period, during regularly scheduled maintenance HD treatment. Each week, enrollees will be introduced to a new skill, all taught in distinctive VR environments-with immersive sessions lasting no more than 30 minutes. The investigators' 5-week positive psychological intervention covers the following topics: (1) noticing positive events, (2) amplifying positive events, (3) gratitude, (4) behavioral activation, (5) mindfulness/meditation, (6) positive reappraisal, (7) personal strengths, and (8) acts of kindness. Delivery of intervention content will require VR immersion for no more than 30 minutes during each HD session (i.e., 30-min. sessions thrice weekly). VR immersion will only occur chairside when patients are already sedentary and in a seated position during regularly scheduled HD treatment, thus avoiding increased sedentarism.
  Interventions: Behavioral: Joviality(TM)
- Inert Virtual Reality (Active Comparator): Participants randomized to the control arm will receive a rigorous placebo following clinical trial guidelines of VR-CORE, which consists of 2-dimensional (2D) non-immersive visual content displayed on the head-mounted display. Footage of wildlife and nature-based settings are visually displayed as part of the 'Sham' VR with inert music that does not promote high levels of relaxation or distraction. The 'Sham' VR experience has very passive features, such that it mimics viewing content on a large flat screen television. Passive viewing during the 'Sham' VR experience rotates content using twenty different videos and has a duration time that is matched to that of JovialityTM over the 5-week intervention period.
  Interventions: Other: Inert Virtual Reality

INTERVENTIONS:
Behavioral: Joviality(TM) — 5-week positive psychological intervention delivered using 3D virtual reality software that is immersive and uses a head-mounted display
  Other Names: Virtual Reality-based Psychotherapy
  Arms: Virtual Reality Treatment
Other: Inert Virtual Reality — Participants randomized to the control arm will receive a rigorous placebo following clinical trial guidelines of VR-CORE, which consists of 2-dimensional (2D) non-immersive visual content displayed on the head-mounted display. Footage of wildlife and nature-based settings are visually displayed as part of the Sham VR with inert music that does not promote high levels of relaxation or distraction.
  Arms: Inert Virtual Reality

SUMMARY:
The long-term goal is to create behavioral health technologies to advance the science that leverages state-of-the-art technology to delivery psychotherapeutic treatment to individuals on hemodialysis (HD) to improve their emotional well-being, quality of life, and overall health. The objective in this small R01 study is to design a virtual reality (VR) platform, that fully immerses users into a fictitious lifelike environment, to deliver an evidence-based positive psychological intervention and to test whether it improves the emotional well-being of individuals on HD with comorbid depression. In this proposed 2-arm randomized controlled trial, the investigators hypothesize that delivery of psychotherapy in individuals on HD using a VR environment will prove feasible and will result in significant improvements in depressive symptoms, quality of life, and treatment adherence, along with reduced rates of hospitalization when compared to an active control condition-all while serving as a cost-effective and far-reaching platform for expansive dissemination.

The Specific Aims are:

Aim #1: To develop VR software to immersively deliver the skills taught in a 5-week evidence-based positive psychological intervention in individuals on HD to improve their emotional well-being.

Aim #2: To evaluate the acceptability and feasibility of a 5-week positive psychological intervention, delivered using a VR platform through consideration of rates of recruitment, refusal, retention, (non)compliance, and adherence.

Aim #3: To test initial efficacy of the VR-based psychotherapeutic intervention, compared to a control arm, on outcomes of depression, psychological well-being, quality of life, treatment adherence, HD sessions missed, and hospitalizations in HD patients.

Knowledge gained from completion of the proposed research will result in the first VR software application to deliver psychotherapy to individuals on HD, while simultaneously allowing them to leave the confines of the clinic and virtually travel to distant regions of the world. This new therapeutic approach can be used to successfully address the added burden of psychological distress experienced by individuals on HD, with the potential to positively impact their quality of life, engagement in healthful behaviors, and overall healthy longevity. And, these findings will yield data essential for a fully-powered trial testing important health outcomes and biomarkers in individuals on HD.

DETAILED DESCRIPTION:
Hemodialysis (HD) is a taxing procedure with extensive illness burden and arduous self-care demands. As such, more than 30% of individuals on HD experience elevated symptoms of depression-and, research shows that comorbid depression is associated with adverse kidney disease outcomes, greater risk of hospitalization, and decreased survival rates. Current interventions to treat depressive symptoms in individuals on HD are resource intensive, infrequently administered, and often involve delivery of psychotherapy by highly-trained clinicians via multiple face-to-face communications. There remains a critical scientific gap for easily disseminatable and efficient strategies to improve emotional well-being profiles of individuals on HD in the U.S. and around the world. The objective in this small R01 study is to design a virtual reality (VR) platform that fully immerses users into a fictitious lifelike environment, to deliver an evidence-based positive psychological intervention and to test whether it improves the emotional well-being of individuals on HD with comorbid depression. For instance, during the module focused on mindfulness/meditation, the investigators will use a head-mounted display to fully immerse and transport individuals on HD to an open field beside a calming stream where they will engage in a 12-minute guided meditation. As such, the investigators propose to conduct a 2-arm randomized controlled trial in which individuals on HD (N=84) will be randomly assigned to receive either the JovialityTM VR-based positive psychological intervention or an active control condition (i.e., 2-dimensional wildlife footage and nature-based settings with inert music). The investigators hypothesize that chairside delivery of psychotherapeutic treatment in individuals on HD using a VR environment will prove feasible and will result in significant improvements in depressive symptoms, quality of life, and treatment adherence, with lower evident rates for missed HD sessions and lower hospitalizations-all while serving as a more cost-effective and far- reaching platform that will greatly expand dissemination. Knowledge gained from completion of the proposed research will result in the first VR software application to deliver psychotherapy to HD patients, while simultaneously allowing them to leave the confines of the clinic and virtually travel to distant regions of the world.

ELIGIBILITY:
Inclusion Criteria:

* 1) HD patient with at least three months since treatment initiation
* 2) Beck Depression Inventory-II (BDI-II) score ≥11
* 3) age 21 or older
* 4) visual and audio acuity to immerse in our VR world
* 5) fluent in English or Spanish

Exclusion Criteria:

* 1) unavailable for study period
* 2) prevalent cognitive impairment denoting dementia
* 3) physical limitation restricting use of a head-mounted display
* 4) history of epilepsy, seizures, or vertigo.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment | Through study completion, an average 6 months.
  Proportion of potential enrollees who were approached for recruitment.
Feasibility: Retention rates | Post-intervention at 6-months
  Defined as completing all post-intervention assessments, categorized as a binary outcome Target: ≥75%
Feasibility: Non-Compliance/Adherence | Immediately post-intervention at 5-weeks
  Measured by the proportion of the intervention completed (e.g., number of virtual reality environments viewed out of the total possible available across skill lessons in the intervention). Target: ≥75%
Feasibility: Refusal rates | Before enrollment
  Proportion of potential enrollees who were approached for recruitment but decided not to enroll.
Acceptability as assessed by whether a participant would recommend the JovialityTM software | Immediately post-intervention at 5-weeks
  Acceptability as measured by whether a participant would recommend JovialityTM to other HD patients (0 definitely not, to 10 definitely yes). Target: ≥8.0

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Depressive symptomatology will be assessed using the Beck Depression Inventory-II. Scores range from 1 to 40 where a higher score indicates worse symptoms of depression.
Kidney Disease and Quality of Life | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Kidney Disease and Quality of Life (KDQOL-SF™). The scoring procedure first transforms the raw precoded numeric values of items to a 0-100 possible range, with higher transformed scores reflecting better quality of life.
Number of missed hemodialysis treatment sessions | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Research staff will extract information from patient medical records to record the number of missed hemodialysis treatment sessions
Emergency department visits and/or hospitalizations | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Research staff will extract information from patient medical records to record the number of emergency department visits and days of hospitalizations.
Patient-Reported Outcomes Measurement Information System (PROMIS) computer adaptive test for depressive symptoms | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) computer adaptive test for depressive symptoms (range values: 28- 140) will serve as an additional measure to triangulate findings of the Beck Depression Inventory-II.
  A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for anxiety | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for anxiety (range values: 29-145) will be used. A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for perceived stress | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for perceived stress (range values: 29-145) will be used.
  A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for life satisfaction | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for life satisfaction (range values: 10-60) will be used. A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for positive affect | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for positive affect (range values: 34-170) will be used.
  A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for life meaning and purpose | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for life meaning and purpose (range values 4-60) will be used. A higher PROMIS T-score represents more of the concept being measured.
Patient-Reported Outcomes Measurement Information System (PROMIS) for self-efficacy for managing emotions in the context of a chronic condition | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The PROMIS adaptive measures for self-efficacy for managing emotions in the context of a chronic condition (range values: 25-125) will be used. A higher PROMIS T-score represents more of the concept being measured.
Psychological well-being measured with the 7-item State Optimism Measure | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Additional measures of psychological well-being will include the optimism using the 7-item State Optimism Measure. Scoring is mean score of items 1-7 with a higher score indicating greater state optimism.
Psychological well-being measured with the Emotional Vitality Measure | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  Additional measures of psychological well-being will also include emotional vitality (range values 0-110), as measured using select items of the General Well-being Schedule. There are three proposed cut-points: total scores of 0-60 reflect "severe distress", 61-72 "moderate distress" and 73-110 "positive well-being"
Psychological well-being measured with the Flourishing Index | Baseline, immediately post-intervention (5-weeks) and at follow-up (3- and 6-months post-intervention)
  The "Flourish" measure is obtained by summing the scores from each of the first five domains. The "Secure Flourish" measure is obtained by summing the scores from all six domains including the financial and material stability domain. Each of the questions is assessed on a scale of 0-10.
  The secure flourishing index score is obtained by summing the scores from the twelve questions in all six domains and results in a score from 0 - 120. Often, for purposes of interpretation, the flourishing and secure flourishing scores are reported as averages of the questions (rather than sums) so that all scores are on a scale of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Hernandez, PhD, Principal Investigator — University of Illinois Urbana-Champaign; Sandraluz Lara-Cinisomo, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (3):
- United States (3):
  - DaVita Little Village Dialysis PD, Chicago, Illinois
  - UI Health - Dialysis Unit, EEI Suite 2028, Chicago, Illinois
  - DaVita Garfield Kidney Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Although the final dataset will be stripped of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of participants with unusual characteristics. Thus, investigators will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to use data only for research purposes and not to identify any individual participant; (2) a commitment to secure the data using appropriate technology; and (3) a commitment to destroy or return data after analyses are completed. If additional outputs result from this research that would be appropriate to share with a wider audience, the investigators will work with the Research Data Service at the University Library to determine appropriate venues for archiving and sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IDP and supporting information described above will be made available no later than 12 months after primary completion date.
Access Criteria: IDP will be shared through data use agreements created and executed by the University of Illinois Urbana Champaign (UIUC).

REFERENCES:
- [Derived] Hernandez R, Wilund K, Solai K, Tamayo D, Fast D, Venkatesan P, Lash JP, Lora CM, Martinez L, Martin Alemany G, Martinez A, Kwon S, Romero D, Browning MHEM, Moskowitz JT. Positive Psychological Intervention Delivered Using Virtual Reality in Patients on Hemodialysis With Comorbid Depression: Protocol and Design for the Joviality Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 16;12:e45100. doi: 10.2196/45100. PMID 37327026